CLINICAL TRIAL: NCT00318773
Title: Short-Term Versus Long-Term Treatment for Severe PMS
Brief Title: Short-Term Versus Long-Term Treatment for Severe Premenstrual Syndrome (PMS)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Ellen W. Freeman, PhD, Research Professor, University of Pennsylvania, Department of Obstetrics/Gynecology
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R01HD018633 (NIH)
Record Dates: First submitted 2006-04-25; First posted 2006-04-27 (Estimated); Last update posted 2009-02-27 (Estimated); Status verified 2006-04

CONDITIONS: Premenstrual Syndrome
Keywords: PMS; PMDD; sertraline; antidepressant; extended treatment; relapse
MeSH Terms: conditions — Premenstrual Syndrome; Recurrence | interventions — Sertraline

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: sertraline — 50 - 100 mg daily for 2 weeks before each menses for 4 months or 12 months and then switched to placebo.

SUMMARY:
Serotonergic antidepressants are clearly effective for premenstrual syndrome (PMS). This study compares short-term treatment (4 months) and long-term treatment (12 months) with sertraline to determine how long medication should be continued after achieving a good response, how soon symptoms return after stopping medication, and whether symptoms are further improved with long-term treatment. Multiple hypotheses include the following: The percent of relapsed subjects is greater with short-term treatment; relapse is swifter with short-term treatment; relapsed subjects improve swiftly when returned to medication; patient satisfactions and quality of life are more improved with long-term treatment.

DETAILED DESCRIPTION:
Severe PMS is a chronic and complex mood disorder that involves mood, behavioral and physical symptoms linked to the menstrual cycle with severity that disrupts functioning for as much as several weeks each menstrual cycle. Estimates indicate that 20-25% of menstruating women experience severe PMS. The efficacy of serotonergic antidepressants is clearly demonstrated for severe forms of PMS in short-term treatment trials. This study compares short-term treatment (4 months) and long-term treatment (12 months) with sertraline in a randomized, placebo-controlled design. The purpose is to determine how long medication should be continued following symptom relief, to what extent and how rapidly symptoms return after stopping medication, and whether there is any additional improvement with long-term treatment.

Following a screen period for 2-3 menstrual cycles that includes a placebo-treated cycle, eligible women are randomized double-blind to the short-term or long-term treatment arm. Subjects are switched (double-blind) to placebo after 4 months or 12 months of sertraline treatment. All subjects continue the study for a total of 21 months and receive either sertraline or the matching placebo in this interval. Subjects whose symptoms return are given open-label sertraline without breaking the study blind. Subjects rate symptoms daily throughout the study using the Penn Daily Symptom Report. Other assessments are conducted at monthly intervals and include the Clinical Global Impressions Rating Scale, Sheehan Disability Scale, Hamilton Depression Rating Scale, Endicott Quality of Life Questionnaire and the Cohen Perceived Stress Scale. The overall duration of the study is expected to be 5-6 years.

ELIGIBILITY:
Inclusion Criteria:

* Women with PMS for at least 1 year.
* Ages 18-45 years
* Regular menstrual cycles in normal range (22-36 days) for at least 6 months
* In general good health as determined by physical examination and blood tests.
* Evidence of ovulation using a urine test.
* Meeting stated criteria for PMS.
* Signed informed consent.

Exclusion Criteria:

* Any prescription, over-the-counter, herbal or non-medical therapies for PMS.
* Use of psychotropic medications that cannot be stopped for the duration of the study.
* Other current psychiatric diagnoses as determined by SCID interview.
* Alcohol or substance abuse/dependence or suicide attempt within the past 12 months; lifetime history of psychosis, bipolar disorder and clearly identifiable severe personality disorder.
* Hysterectomy, symptomatic endometriosis, irregular menstrual cycles,any severe or unstable medical illness.
* Lack of medically-approved contraception, currently pregnant, intention to become pregnant or breast feeding.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 174 (Actual)
Dates: Start 2002-02; Primary Completion 2007-12 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Penn Daily Symptom Report (DSR) | daily

SECONDARY OUTCOMES:
Hamilton Depression Scale | monthly
Quality of Life Questionnaire | monthly
Sheehan Disability Scales | monthly
Clinical Global Rating of Severity and Improvement | monthly

CONTACTS AND LOCATIONS:
Overall Officials: Ellen W Freeman, PhD, Principal Investigator — University of Pennsylvania, School of Medicine, Department of Ob/Gyn; Steven J Sondheimer, MD, Principal Investigator — University of Pennsylvania; Karl Rickels, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Department of Obstetrics/Gynecology, University of Pennsylvania, School of Medicine, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Freeman EW, Rickels K, Sammel MD, Lin H, Sondheimer SJ. Time to relapse after short- or long-term treatment of severe premenstrual syndrome with sertraline. Arch Gen Psychiatry. 2009 May;66(5):537-44. doi: 10.1001/archgenpsychiatry.2008.547. PMID 19414713